CLINICAL TRIAL: NCT02582814
Title: A Clinical Pharmacology and Long Term Study to Evaluate the Safety, Efficacy, Pharmacokinetics and Pharmacodynamics of Dapagliflozin Therapy in Combination With Insulin in Japanese Subjects With Type 1 Diabetes Who Have Inadequate Glycemic Control
Brief Title: The Safety and Efficacy of Dapagliflozin Therapy in Combination With Insulin in Japanese Subjects With T1DM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D1695C00001
Record Dates: First submitted 2015-10-20; First posted 2015-10-21 (Estimated); Results first posted 2019-04-12 (Actual); Last update posted 2019-04-12 (Actual); Status verified 2019-01

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Japanese patients with type 1 diabetes with inadequate glycemic control on insulin
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — dapagliflozin

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: No

ARMS (2):
- dapagliflozin 5mg + insulin (Experimental): dapagliflozin tablet 5mg + adjustable insulin
  Interventions: Drug: Dapagliflozin 5 mg
- dapagliflozin 10mg + insulin (Experimental): dapagliflozin tablet 10mg + adjustable insulin
  Interventions: Drug: Dapagliflozin 10mg

INTERVENTIONS:
Drug: Dapagliflozin 5 mg — Dapagliflozin, a blood glucose lowering drug. Oral dose
  Arms: dapagliflozin 5mg + insulin
Drug: Dapagliflozin 10mg — Dapagliflozin, a blood glucose lowering drug. Oral dose
  Arms: dapagliflozin 10mg + insulin

SUMMARY:
This study will enroll eligible subjects into a long-term safety study (Part B).

Japanese male and female patients with T1DM and age 18 to 75 years, with inadequate glycemic control on insulin defined as HbA1c ≥ 7.5% and ≤ 10.5% at screening visit. As a condition of enrollment, subjects must be on a total daily insulin dose of ≥ 0.3 U/kg/day for at least 3 months prior to the screening visit. The study design of Part B is a randomized, open-label, 2 arm, parallel-group design. 140 Japanese subjects in total will be randomized in a 1:1 ratio into one of the two treatment arms; dapagliflozin 5 mg or dapagliflozin 10 mg.

ELIGIBILITY:
Inclusion Criteria:

* Signed Written Informed Consent
* Diagnosis of T1DM. In addition, the following criteria also needs to be met; Central laboratory test of C-peptide < 0.7 ng/mL
* Insulin use for at least 12 months prior to the enrolment per subject report or medical records and Method of insulin administration (MDI or CSII) must have been unchanged for at least 3 months prior to the enrolment per subject report or medical records. Subjects must be taking a total daily insulin dose of ≥ 0.3 U/kg/day for at least 3 months prior to the enrolment. If on MDI insulin administration subject must be on ≥ 3x injections per day.
* Japanese men and women
* Screening Visit: Central laboratory HbA1c ≥ 7.5% and ≤ 10.5%
* BMI ≥ 20.0 kg/m² at visit 1
* Age 18 to 75 years, inclusive

Exclusion Criteria:

- Target Disease Exceptions History of T2DM Maturity onset diabetes of young (MODY) Any anti-hyperglycemic agent use, other than α-GI or insulin, within 1 month prior to the enrolment.

Use of thiazolidinediones within 6 months prior to the enrolment History of DKA requiring medical intervention within 1 month prior to the enrolment History of hospital admission for glycemic control (either hyperglycemia or hypoglycemia) within 1 month prior to the enrolment

* Medical History and Concurrent Diseases Malignancy within 5 years of the enrolment (with the exception of treated basal cell or treated squamous cell carcinoma) History of bladder cancer History of radiation therapy to the lower abdomen or pelvis at any time
* Physical and Laboratory Test Findings Aspartate aminotransferase (AST) > 3x upper limit of normal (ULN) Alanine aminotransferase (ALT) > 3x ULN Serum total bilirubin (TB) > 2.0 mg/dL (34.2 μmol/L) Estimated GFR (eGFR) by the Japanese Society of Nephrology formula ≤ 45 mL/min/1.73m2 Hemoglobin ≤ 11.0 g/dL (110 g/L) for men; hemoglobin ≤ 10.0 g/dL (100 g/L) for women.

Positive for hepatitis B surface antigen or anti-hepatitis C virus antibody Abnormal Free T4

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2015-10-26 (Actual); Primary Completion 2017-06-15 (Actual); Study Completion 2017-06-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (24):
- Japan (24):
  - Research Site, Aizu Wakamatsu-shi
  - Research Site, Chūōku
  - Research Site, Fukuoka
  - Research Site, Fukuyama-shi
  - Research Site, Funabashi-shi
  - Research Site, Hamamatsu
  - Research Site, Hirosaki-shi
  - Research Site, Ise-shi
  - Research Site, Kagoshima
  - Research Site, Koriyama-shi
  - Research Site, Kumamoto
  - Research Site, Kunitachi-shi
  - Research Site, Minatoku
  - Research Site, Nagoya
  - Research Site, Oyama-shi
  - Research Site, Ōita
  - Research Site, Ōtsu
  - Research Site, Sapporo
  - Research Site, Sendai
  - Research Site, Shinjyuku-ku
  - Research Site, Suita-shi
  - Research Site, Tama-shi
  - Research Site, Tsukuba
  - Research Site, Yokohama

REFERENCES:
- See also: D1695C00001_SAP_redacted — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=3797&filename=D1695C00001_SAP_Redacted.pdf
- See also: D1695C00001_CSP_redacted — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=3797&filename=D1695C00001_CSP_redacted.pdf

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dapagliflozin 5mg + Insulin | Dapagliflozin 10mg + Insulin
Started | 76 | 75
Completed | 67 | 68
Not Completed | 9 | 7
Not completed — Study-specific withdrawal criteria | 1 | 0
Not completed — Withdrawal by Subject | 4 | 3
Not completed — Adverse Event | 4 | 4

BASELINE CHARACTERISTICS:
Population: Randomized set
Groups:
- Total: Total of all reporting groups
Arm/Group | Dapagliflozin 5mg + Insulin | Dapagliflozin 10mg + Insulin | Total
Number analyzed (Participants) | 76 | 75 | 151
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.7 (12.85) | 48.9 (12.93) | 48.3 (12.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 42 | 75
  Male | 43 | 33 | 76
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 76 | 75 | 151
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] | 25.28 (3.635) | 24.66 (2.806) | 24.97 (3.254)
Duration of T1DM [Mean (Standard Deviation); unit: years] | 14.60 (8.420) | 15.94 (10.328) | 15.27 (9.409)
HbA1c [Mean (Standard Deviation); unit: Percent] | 8.43 (0.711) | 8.40 (0.715) | 8.42 (0.711)
C-peptide [Count of Participants; unit: Participants]
  < 0.1 ng/mL | 63 | 65 | 128
  >= 0.1 ng/mL | 13 | 10 | 23

OUTCOME MEASURES:

1. Primary Outcome: Overall Adverse Event Summary
Description: To evaluate safety and tolerability of long-term treatment (52 weeks) of dapagliflozin 5mg and 10 mg in Japanese patients with T1DM with inadequate glycemic control under standard insulin therapy.
Time Frame: From baseline to 52 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Dapagliflozin 5mg + Insulin | Dapagliflozin 10mg + Insulin
Number analyzed (Participants) | 76 | 75
Participants
  Adverse Events: At least one events | 67 | 55
  Related Adverse Events: At least one events | 23 | 22
  SAE: At least one events | 7 | 3
  AEs leading to discontinuation: At least one events | 4 | 4
  Death: At least one events | 0 | 0

2. Primary Outcome: Hypoglycemia
Description: as for outcome 1
Time Frame: From baseline to 52 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Dapagliflozin 5mg + Insulin | Dapagliflozin 10mg + Insulin
Number analyzed (Participants) | 76 | 75
Participants
  Any Hypoglycemia Episodes: At least one events | 75 | 75
  Severe Hypoglycemia: At least one events | 2 | 5
  Documented Symptomatic Hypoglycemia: At least one events | 67 | 73
  Asymptomatic Hypoglycemia: At least one events | 60 | 64
  Probable Symptomatic Hypoglycemia: At least one events | 13 | 14
  Relative Hypoglycemia: At least one events | 14 | 11

3. Primary Outcome: Diabetic Ketoacidosis (DKA)
Description: as for outcome 1
Time Frame: From baseline to 52 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Dapagliflozin 5mg + Insulin | Dapagliflozin 10mg + Insulin
Number analyzed (Participants) | 76 | 75
Participants
  Definite DKA: At least one events | 2 | 1
  Possible DKA: At least one events | 1 | 0
  Unlikely DKA: At least one events | 0 | 0

4. Secondary Outcome: Adjusted Change From Baseline in HbA1c
Description: To assess the efficacy of long-term treatment (24/52 weeks) of dapagliflozin 5mg and 10 mg in Japanese patients with T1DM inadequately controlled on insulin therapy.
Time Frame: From baseline to 24/52 weeks
Population: All available post-baseline data were included in analysis. Nubmer of observations at each time point is presented in the table below.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent
Arm/Group | Dapagliflozin 5mg + Insulin | Dapagliflozin 10mg + Insulin
Number analyzed (Participants) | 74 | 74
percent
  Week 24: number analyzed (Participants) | 72 | 72
  Week 24 | -0.52 [-0.66 to -0.38] | -0.66 [-0.80 to -0.53]
  Week 52: number analyzed (Participants) | 68 | 68
  Week 52 | -0.33 [-0.50 to -0.15] | -0.36 [-0.53 to -0.18]

5. Secondary Outcome: Adjusted Percent Change From Baseline in Total Daily Insulin Dose
Description: as for outcome 4
Time Frame: From baseline to 24/52 weeks
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Dapagliflozin 5mg + Insulin | Dapagliflozin 10mg + Insulin
Number analyzed (Participants) | 73 | 73
percent change
  Week 24: number analyzed (Participants) | 72 | 71
  Week 24 | -15.30 [-18.55 to -11.92] | -15.14 [-18.43 to -11.73]
  Week 52: number analyzed (Participants) | 69 | 68
  Week 52 | -12.27 [-15.92 to -8.46] | -13.13 [-16.77 to -9.33]

6. Secondary Outcome: Adjusted Percent Change From Baseline in Body Weight
Description: as for outcome 4
Time Frame: From baseline to 24/52 weeks
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Dapagliflozin 5mg + Insulin | Dapagliflozin 10mg + Insulin
Number analyzed (Participants) | 74 | 74
percent change
  Week 24: number analyzed (Participants) | 72 | 72
  Week 24 | -3.88 [-4.74 to -3.02] | -5.26 [-6.11 to -4.41]
  Week 52: number analyzed (Participants) | 68 | 68
  Week 52 | -4.25 [-5.29 to -3.21] | -5.96 [-6.98 to -4.93]

7. Secondary Outcome: Adjusted Change From Baseline in Glycoalbumin
Description: as for outcome 4
Time Frame: From baseline to 24/52 weeks
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: percent
Arm/Group | Dapagliflozin 5mg + Insulin | Dapagliflozin 10mg + Insulin
Number analyzed (Participants) | 74 | 74
percent
  Week 24: number analyzed (Participants) | 72 | 72
  Week 24 | -2.26 [-2.83 to -1.70] | -2.63 [-3.22 to -2.04]
  Week 52: number analyzed (Participants) | 68 | 68
  Week 52 | -1.49 [-2.18 to -0.77] | -1.68 [-2.41 to -0.96]

8. Secondary Outcome: Adjusted Change From Baseline in Average Daily Glucose Measured by 6-point SMBG
Description: as for outcome 4
Time Frame: From baseline to 24/52 weeks
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Dapagliflozin 5mg + Insulin | Dapagliflozin 10mg + Insulin
Number analyzed (Participants) | 73 | 72
mg/dL
  Week 24: number analyzed (Participants) | 72 | 70
  Week 24 | -9.37 [-15.80 to -2.94] | -15.06 [-21.62 to -8.51]
  Week 52: number analyzed (Participants) | 67 | 67
  Week 52 | -11.62 [-18.62 to -4.62] | -12.93 [-19.99 to -5.88]

9. Secondary Outcome: Adjusted Change From Baseline in Post-prandial Glucose Measured by 6-point SMBG
Description: as for outcome 4
Time Frame: From baseline to 24/52 weeks
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Dapagliflozin 5mg + Insulin | Dapagliflozin 10mg + Insulin
Number analyzed (Participants) | 73 | 73
mg/dL
  Week 24: number analyzed (Participants) | 72 | 71
  Week 24 | -2.33 [-11.18 to 6.51] | -10.08 [-19.04 to -1.12]
  Week 52: number analyzed (Participants) | 67 | 68
  Week 52 | -6.40 [-15.45 to 2.64] | -5.24 [-14.32 to 3.83]

10. Secondary Outcome: Proportion of Subjects Achieving HbA1c Reduction of 0.5 Percent Without Severe Hypoglycemia
Description: To assess the efficacy of long-term treatment (24/52 weeks) of dapagliflozin 5mg and 10 mg in Japanese patients with T1DM inadequately controlled on insulin
Time Frame: From baseline to 24/52 weeks
Population: Subjects with non-missing HbA1c baseline and Week24/52 (LOCF) values were included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dapagliflozin 5mg + Insulin | Dapagliflozin 10mg + Insulin
Number analyzed (Participants) | 74 | 75
percentage of participants
  Week 24 | 60.8 [48.8 to 72.0] | 61.3 [49.4 to 72.4]
  Week 52 | 51.4 [39.4 to 63.1] | 41.3 [30.1 to 53.3]

11. Secondary Outcome: Proportion of Subjects Achieving HbA1c Reduction of 0.5 Percent
Description: as for outcome 10
Time Frame: From baseline to 24/52 weeks
Population: Subjects with non-missing HbA1c baseline and Week24/52 (LOCF) values were included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dapagliflozin 5mg + Insulin | Dapagliflozin 10mg + Insulin
Number analyzed (Participants) | 74 | 75
percentage of participants
  Week 24 | 62.2 [50.1 to 73.2] | 66.7 [54.8 to 77.1]
  Week 52 | 51.4 [39.4 to 63.1] | 45.3 [33.8 to 57.3]

12. Secondary Outcome: Proportion of Subjects Achieving HbA1c < 7.0 Percent
Description: as for outcome 10
Time Frame: From baseline to 24/52 weeks
Population: Subjects with non-missing HbA1c baseline and Week24/52 (LOCF) values were included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dapagliflozin 5mg + Insulin | Dapagliflozin 10mg + Insulin
Number analyzed (Participants) | 74 | 75
percentage of participants
  Week 24 | 9.5 [3.9 to 18.5] | 5.3 [1.5 to 13.1]
  Week 52 | 6.8 [2.2 to 15.1] | 2.7 [0.3 to 9.3]

13. Secondary Outcome: Adjusted Change From Baseline in SBP in Subjects With Baseline SBP/DBP >= 140/90 mmHg
Description: as for outcome 10
Time Frame: From baseline to 24/52 weeks
Population: Subjects with baseline SBP >= 140mmHg and/or baselien DBP >= 90mmHg were included in analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Dapagliflozin 5mg + Insulin | Dapagliflozin 10mg + Insulin
Number analyzed (Participants) | 19 | 13
mmHg
  Week 24: number analyzed (Participants) | 19 | 12
  Week 24 | -5.8 [-11.2 to -0.3] | -12.0 [-19.0 to -5.0]
  Week 52: number analyzed (Participants) | 18 | 12
  Week 52 | -9.8 [-15.1 to -4.5] | -14.2 [-20.7 to -7.6]

14. Primary Outcome: Vital Signs (Heart Rate)
Description: as for outcome 1
Time Frame: From baseline to 52 weeks
Population: Subjects with both non-missing baseline and non-missing Week 52 were included.
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Dapagliflozin 5mg + Insulin | Dapagliflozin 10mg + Insulin
Number analyzed (Participants) | 76 | 75
bpm | -0.3 (10.07) | 0.4 (8.89)

15. Primary Outcome: ECGs
Description: as for outcome 1
Time Frame: From baseline to 52 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Dapagliflozin 5mg + Insulin | Dapagliflozin 10mg + Insulin
Number analyzed (Participants) | 76 | 75
Participants
  Baseline: NORMAL | 65 | 67
  Baseline: ABNORMAL | 11 | 8
  Baseline: NOT REPORTED | 0 | 0
  Week 52: NORMAL | 69 | 67
  Week 52: ABNORMAL | 5 | 8
  Week 52: NOT REPORTED | 2 | 0

16. Primary Outcome: Clinical Laboratory Measures, Urine Test Results (Any Marked Abnormality)
Description: as for outcome 1
Time Frame: From baseline to 52 weeks
Population: Subjects with non-missing post-baseilne measurements were included.
Measure: Count of Participants; unit: Participants
Arm/Group | Dapagliflozin 5mg + Insulin | Dapagliflozin 10mg + Insulin
Number analyzed (Participants) | 76 | 75
Participants
  Hematocrit (> 55%): number analyzed (Participants) | 74 | 75
  Hematocrit (> 55%) | 1 | 0
  Hemoglobin (> 18g/dL) | 2 | 1
  Creatinine (>1.5 x ULN pre Rx) | 0 | 1
  Creatin kinase (> 5x ULN) | 1 | 1
  Bicarbonate (<= 13 mEq/L) | 1 | 0
  P (<=1.8/2.1mg/dL for age<=/>65) | 1 | 1
  UACR (> 1800mg/g) | 0 | 1

17. Primary Outcome: Vital Signs (Blood Pressure)
Description: as for outcome 1
Time Frame: From baseline to 52 weeks
Population: Subjects with both non-missing baseline and non-missing Week 52 were included.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Dapagliflozin 5mg + Insulin | Dapagliflozin 10mg + Insulin
Number analyzed (Participants) | 76 | 75
mmHg
  Change from baseline in SBP(mmHg) at Week 52: number analyzed (Participants) | 68 | 68
  Change from baseline in SBP(mmHg) at Week 52 | -3.4 (11.41) | -2.9 (12.55)
  Change from baseline in DBP(mmHg) at Week 52: number analyzed (Participants) | 68 | 68
  Change from baseline in DBP(mmHg) at Week 52 | -0.6 (8.21) | -1.0 (7.89)

ADVERSE EVENTS:
Time Frame: 1 year. Non-serious adverse event (AE): onset on or after the 1st day of dose up to on or prior to the last day of dose plus 4 days. Serious AE: onset on or after the 1st day of dose up to on or prior to the last day of dose plus 30 days
Description: Only hypoglycemia/ DKA reported as a serious adverse event are included.
Arm/Group | Dapagliflozin 5mg + Insulin | Dapagliflozin 10mg + Insulin
All-Cause Mortality (participants affected / at risk) | 0/76 | 0/75
Serious Adverse Events (participants affected / at risk) | 7/76 | 3/75
Other Adverse Events (participants affected / at risk) | 66/76 | 55/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dapagliflozin 5mg + Insulin (N=76) | Dapagliflozin 10mg + Insulin (N=75)
VITREOUS HAEMORRHAGE (Eye disorders) | 0 (0) | 1 (1)
COLITIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
DIABETIC KETOACIDOSIS (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
HYPOGLYCAEMIC COMA (Nervous system disorders) | 0 (0) | 1 (1)
ATRIAL FIBRILLATION (Cardiac disorders) | 1 (1) | 0 (0)
HEPATIC FUNCTION ABNORMAL (Hepatobiliary disorders) | 1 (1) | 0 (0)
GASTROENTERITIS (Infections and infestations) | 1 (1) | 0 (0)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
ABORTION SPONTANEOUS (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dapagliflozin 5mg + Insulin (N=76) | Dapagliflozin 10mg + Insulin (N=75)
NASOPHARYNGITIS (Infections and infestations) | 25 (39) | 32 (44)
PHARYNGITIS (Infections and infestations) | 5 (6) | 9 (13)
GASTROENTERITIS (Infections and infestations) | 7 (8) | 8 (10)
DENTAL CARIES (Gastrointestinal disorders) | 0 (0) | 5 (5)
ECZEMA (Skin and subcutaneous tissue disorders) | 4 (4) | 4 (4)
THIRST (General disorders) | 4 (4) | 4 (4)
HEADACHE (Nervous system disorders) | 4 (4) | 6 (12)
POLLAKIURIA (Renal and urinary disorders) | 7 (7) | 6 (6)
KETOSIS (Metabolism and nutrition disorders) | 4 (8) | 7 (15)
BRONCHITIS (Infections and infestations) | 2 (5) | 4 (4)
INFLUENZA (Infections and infestations) | 4 (4) | 2 (2)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 6 (9) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-03-16): https://cdn.clinicaltrials.gov/large-docs/14/NCT02582814/SAP_000.pdf
  • Study Protocol (2016-12-14): https://cdn.clinicaltrials.gov/large-docs/14/NCT02582814/Prot_001.pdf